CLINICAL TRIAL: NCT04895839
Title: PC-PEP Phase 4: Predictors of Mental Health in Men With Prostate Cancer Undergoing a Patient Empowerment Program
Brief Title: Predictors of Mental Health in Men With Prostate Cancer Undergoing a Patient Empowerment Program
Acronym: PC-PEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriela Ilie (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor-Investigator, Gabriela Ilie, Faculty/Assistant Professor, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PC_PEP_Phase 4_Protocol
Record Dates: First submitted 2021-05-13; First posted 2021-05-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: mental health; quality of life; empowerment program
MeSH Terms: conditions — Prostatic Neoplasms; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental)
  Interventions: Behavioral: Patient Empowerment Program

INTERVENTIONS:
Behavioral: Patient Empowerment Program — The 6 months "at home" program focuses on aerobic and strength training, pelvic floor muscle exercises, meditation, social connection, and overall healthy lifestyle practices supported with daily text message/email reminders. The aerobic (5 times/week) and strength (2 times/week) program will comprise of a single 30-minute session daily and will be individualized to each participant. Pelvic floor muscle training will include three, 10-minute sessions and mediation for 10 minutes daily. Intimacy and Connection component of PC-PEP consists of engaging in at least one form of intimacy practice prescribed, per day. Social connection will be fostered by pairing participants up with peers from the study. To encourage program compliance, study participants will receive 3 daily reminders to do their pelvic floor muscle exercises per day plus an additional motivational email daily containing helpful tips.

SUMMARY:
Each year over 20,000 men are diagnosed with prostate cancer in Canada with the majority undergoing some form of treatment option. Radical prostatectomy and/or radiation therapy are common procedures that are effective in the treatment of prostate cancer. However, they typically incur both short- and long-term side effects (e.g. urinary incontinence, sexual dysfunction, reduced physical function, etc) that can negatively impact one's quality of life. This program of research aims to address the most critical needs of PC survivors: the development and evaluation of interventions to address the quality of life impact of PC. This study will test the Prostate Cancer Patient Empowerment Program (PC-PEP) in 400 men, a comprehensive intervention aimed at educating and teaching the men life skills/habits in order to improve their mental health issues, fitness levels and overall quality of life, and to decrease treatment related side effects. The program also aims to improve the overall health of the participants in the long term.

DETAILED DESCRIPTION:
In a survey study of almost 400 survivors of prostate cancer (PC), the investigators found that 17% of them suffered currently from mental health issues, and most were not on medication to address this issue. Compounding issues included urinary and sexual disfunction, poor attendance to support groups, intimacy, problems sleeping and other health problems. To address these many issues directly, with the endorsement of physicians and patients attending our regional PC integrative care conference (April 2018) and expanding on pre-habitation (pre-surgery) science, the investigators created a Patient Empowerment Program (PEP) to be delivered from day one of diagnosis, to educate and teach the men and partners life skills/habits which are aimed to improve their fitness levels and quality of life, and to decrease treatment related side effects. This program is in line with the Auditor General of Nova Scotia's 2017 report endorsing the use of bottom-up evidence-based interventions, created from actively engaging patients in development and process. The investigators aim to trial PC-PEP for men undergoing curative treatment for PC versus a control group receiving standard care. The PC-PEP program includes in-person and multimedia informational, physical activity, pelvic floor, stress reduction, and relationship/connection training. The men are connected with other participants to increase social support and maximize compliance. Technology is used to deliver daily alerts to patients to remind them to engage in the program. A PC-PEP feasibility study of 30 men, over 28 days, showed that the program is feasible, leads to positive outcomes in patients and is highly (9.79/10) endorsed by patients. It is predicted that PC-PEP will improve mental health (primary outcome) and other quality of life outcomes of patients compared with 'usual care'.

A randomized, wait-list controlled clinical trial for men newly diagnosed with PC is currently underway. This next phase will open the program to more men and expand the inclusion criteria. Participants in the PC-PEP will receive the intervention for six months. Introducing a comprehensive empowerment program from day one of diagnosis may mitigate against the high levels of mental distress, short and long-term, suffered by hundreds of Nova Scotian men undergoing curative PC treatment every year, and the burden that treatment related side effects will place on our health care system. Given that the study has the endorsement of patients, clinicians and administrators at Nova Scotia Health, if proven successful it will have the evidence base needed to change the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* History of a prostate cancer diagnosis
* Safe to exercise and do strength training (participants who have recovered from a minor stroke or heart condition in the past will require approval from their Family Physician or Cardiologist to participate in the study. Participants with advanced prostate cancer will need approval from the Study Physician or their Urologist or Oncologist to participate)
* Existing (or willingness to create) email account
* Willingness to access and use daily email and/or text messages
* Ability to follow website links to watch YouTube videos
* Ability to understand and speak English
* Ability to participate in low to moderate levels of physical activity
* Ability and willingness to fill out an online survey at baseline, and 6, 12 and 24 months, and a weekly compliance survey for the six months of the program.
* Deemed to have an expected survival greater than 2 years

Exclusion Criteria:

* Patients deemed unfit to participate in low level exercise eg. including but not limited to a myocardial infarction or stroke within the last year, without approval from their Family Physician or Cardiologist that they are safe to exercise.
* Unable to access the internet and lack of a computer or cellphone to receive emails required for study intervention, or unable to click on a link to successfully watch a YouTube video.
* Men with a predicted survival less than 2 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2130 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Mental Health | 6 - 24 months
  Kessler 10 - assessment of psychological distress. Measured through on-line survey.

SECONDARY OUTCOMES:
General Health (Physical and Mental) Quality of Life as assessed by the 12-item Short Form Health Survey (SF-12) | 6 - 24 months
  The scale has a score range of 0 to 100, with a higher score indicating a better outcome, and a score of 50 indicating the U.S. population average.
Disease Specific Health-Related Quality of Life as assessed by the Functional Assessment of Cancer Therapy-Prostate (FACT-P) | 6 - 24 months
  A 39-item questionnaire. The scale has a total score range of 0-156 with a higher score indicating better quality of life.
Urinary, Bowel, Hormonal, and Sexual Function as assessed by the Expanded Prostate Cancer Index Composite (EPIC) | 6 - 24 months
  A 50-item questionnaire to evaluate patient function and bother after prostate cancer treatment. The scale has a score range of 0-100 with a higher score indicating a better outcome.
Urinary Bother as assessed by the International Prostate Symptom Score (IPSS) | 6 - 24 months
  A 7-item questionnaire. The scale has a score range of 0-35 with a higher score indicating more severe urinary bother.
Health Care Utilization | 6 - 24 months
  This will be assessed through the following survey questions:
  1. During the PAST 6 MONTHS, how many TIMES did you visit a doctor or health care provider for physical illness? (do not include visits while you were in the hospital for your Prostate Cancer treatment (e.g., radiation, surgery, etc)?
  2. During the PAST 6 MONTHS, how many TIMES did you visit a doctor or health care provider for a mental health issue?
  3. How many TIMES did you visit the emergency room in the PAST 6 MONTHS but were not admitted overnight?
  4. How many TIMES were you admitted to the hospital overnight in the PAST 6 MONTHS?
Relationship Satisfaction as assessed by the Dyadic Adjustment Scale (DAS) | 6 - 24 months
  DAS is a 32-item questionnaire that measures an individual's perceptions of their relationship with an intimate partner. The scale has a total score range of 1-151 with a higher score indicating better satisfaction.
Diet as assessed by the Starting the Conversation (STC) Questionnaire | 6 - 24 months
  STC is an 8-item simplified food frequency instrument designed for use in primary care and health-promotion settings. The instrument has a score range of 0-16 with a higher score indicating worse diet.
Sleep Quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | 6 - 24 months
  PSQI included 19self-rated items that assess sleep quality and disturbances over a 1-month time interval. The scale has a score range of 0-21, with a higher score indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (6):
  - Dianne and Irving Kipnes Urology Centre, Edmonton, Alberta
  - BC Cancer - Kelowna (Sindi Ahluwalia Hawkins Centre), Kelowna, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Mount Sinai Hospital, Toronto, Ontario
  - Saskatoon Health Authority, Saskatoon, Saskatchewan
- Prostate Cancer Foundation of New Zealand, Auckland, New Zealand